CLINICAL TRIAL: NCT07368010
Title: End-of-life Care in Mechanically Ventilated Patients: Impact of a Comprehensive Training to Palliative Care in the Intensive Care Setting. A Multicenter Cluster Randomised Trial
Brief Title: End-of-life Care in Mechanically Ventilated Patients: Impact of a Comprehensive Palliative Care Protocol in the Intensive Care Setting
Acronym: ARREVE-3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: University of Burgundy (Other); Centre Hospitalier Universitaire de Saint Louis APHP (Unknown); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC24_0575
Record Dates: First submitted 2025-12-19; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Palliative Care; Withdrawal of Life Support; Intensive Care Medicine; Sedation; Dying Process
Keywords: End of life; intensive care medicine; mechanical ventilation; organ support; withdrawal; life support; sedation; palliative care
MeSH Terms: conditions — Death | interventions — Clinical Protocols; Palliative Care

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative care protocol (Experimental): Protocol for life-support withdrawal and palliative care during the withdrawal process
  Interventions: Other: Protocol for palliative care and life-support withdrawal
- Usual Care (No Intervention): Withdrawal of life support at the end of life will be performed according to the usual practices of the participating ICUs

INTERVENTIONS:
Other: Protocol for palliative care and life-support withdrawal — In the intervention group, end-of-life care will be provided in accordance with the study protocol, which specifies pharmacological management, nursing care, management of life-sustaining organ support, procedures for the assessment of comfort and pain, and support for relatives. Medical and nursing staff in intervention centers will receive on-site, face-to-face training on the care protocol within each ICU. An instructional video detailing the protocol will also be available.
  Arms: Palliative care protocol

SUMMARY:
The ARREVE-3 trial will evaluate whether a structured palliative care protocol can improve end-of-life management for mechanically ventilated ICU patients in whom a decision to withdraw life-sustaining therapies has been made. This cluster-randomized controlled trial compares protocol-based care with usual practice across participating centers. The intervention includes comprehensive guidance on symptom management, sedation, nursing care, withdrawal procedures, and family support, supported by standardized staff training. The primary endpoint is adherence to recommended end-of-life practices, while secondary outcomes assess patient comfort, communication with relatives, and the impact on families and healthcare professionals

DETAILED DESCRIPTION:
Among ICU patients who die after a decision to withdraw life-sustaining therapies, most are receiving mechanical ventilation (MV). Withdrawal of MV may cause discomfort, and end-of-life practices can have a lasting impact on both families and healthcare professionals. Despite international guidelines and recent legislative changes in France, end-of-life practices in the ICU remain highly variable, indicating substantial opportunities for improvement in patient comfort-focused management.

The ARREVE-3 trial aimes to determine whether a structured palliative care protocol for mechanically ventilated patients undergoing withdrawal of life-sustaining therapies improves the quality of the dying process. Developed in collaboration with palliative care specialists, a psychologist, and a sociologist, the protocol provides standardized guidance on pharmacological and non-pharmacological interventions, including symptom assessment tools, sedation strategies, nursing care, and procedures for withdrawal of life-sustaining treatment. Structured recommendations for support of relatives are also included.

ARREVE-3 is a pragmatic, interventional, cluster-randomized controlled trial, with participating ICUs being unit of randomization to minimize contamination between study arms. ICUs randomized to the intervention arm will apply the palliative care protocol, whereas control ICUs will continue to follow usual care. Physicians and nurses in intervention ICUs will receive standardized training from the coordinating team, complemented by a video-based educational module. Designated local champions within each ICU will support implementation and adherence.to the protocol.

The primary endpoint is adherence to the protocol for end-of-life care. Secondary outcomes include patient comfort, quality of communication with relatives, and the impact of the end-of-life process on relatives and healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Patient:

  * Age ≥ 18 years
  * ICU admission for more than 48 hours
  * Receiving invasive mechanical ventilation
  * A documented decision to withdraw life-sustaining therapies, made through a multidisciplinary collegial process and communicated to the designated surrogate decision-maker, family, or relatives
  * At least one visit from a relative prior to the decision to withdraw life-sustaining therapies
  * Provision of informed consent for study participation, or, if the patient lacks decision-making capacity, consent obtained from a relative or legally authorized representative
* Relative:

  * Age ≥ 18 years
  * Has received at least one medical update regarding the patient's clinical status from an ICU physician prior to the decision to withdraw life-sustaining therapies
  * Has provided informed consent for study participation

Exclusion Criteria:

* Patient:

  * Presence of a tracheostomy
  * Brain death or involvement in an organ donation procedure
  * Absence of any visit from a relative
  * Subject to legal guardianship or other legal protection measures
  * Incarcerated patient
  * Participation in another interventional research study focused on end-of-life care
  * Pregnant or breastfeeding woman
* Relative:

  * Inability to understand or speak French
  * Subject to legal guardianship or other legal protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2028-01-10 (Estimated); Study Completion 2029-01-10 (Estimated)

PRIMARY OUTCOMES:
To assess whether, compared with usual care, the implementation of a palliative care protocol for mechanically ventilated patients-combined with dedicated staff training-improves adherence to guidelines. | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients receiving adequate sedation (RASS-5 within one hour before withdrawal of life-sustaining therapies) and withdrawal of mechanical ventilation

SECONDARY OUTCOMES:
Evaluation of Sedation | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Maximum rate of continuous infusion of each sedative agent administered (within 1 hour before the first withdrawal of life sustaining therapies and death)
Evaluation of Sedation | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Number of sedative boluses and number of dose escalations of continuous sedation between inclusion and death
Proportion of Patients Receiving Medications Other Than Sedatives | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients receiving neuromuscular blocking agents, scopolamine, paracetamol (acetaminophen), or antiemetic agents.
Administration of neuromuscular blocking agents | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients receiving neuromuscular blocking agents
Administration of scopolamine | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients receiving scopolamine
Administration of paracetamol (acetaminophen) | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients receiving paracetamol (acetaminophen)
Administration of Receiving antiemetic agents | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients receiving antiemetic agents
The Semi-Lateral (¾ Lateral) Position | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients positioned in the semi-lateral (¾ lateral) position 1 hour before treatment withdrawal and 1 hour before death
Life-Sustaining Organ Support Management | From inclusion to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients receiving dialysis, vasoactive drug and/or ECMO at inclusion and at death
Life-Sustaining Organ Support Management | From inclusion to death, assessed up to 28 days
  Proportion of patients in whom all life-sustaining therapies are discontinued before death
Life-Sustaining Organ Support Management | From inclusion to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients in whom all life-sustaining therapies are withdrawn concomitantly
Life-Sustaining Organ Support Management | From inclusion to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients whith immediate extubation
Time from Inclusion to Extubation | From inclusion to date of extubation, assessed up to 28 days
  Time interval between inclusion and extubation
Assessment of Sedation | From inclusion to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients with a Richmond Agitation-Sedation Scale (RASS) score of -5 or > -4 (≥ -3) 1 hour before withdrawal of the first life-sustaining therapy (mechanical ventilation, vasopressors, or ECMO) and 1 hour before extubation
Assessment of Pain Management | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Higher Behavioral Pain Scale (BPS) score 1 hour before withdrawal of the first life-sustaining therapy (mechanical ventilation, vasopressors, or ECMO); BPS min = 3, max = 12; Higher scores correlate with increased pain intensity.
Assessment of Comfort Management | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients with airway secretion scores of 3 or 4
Assessment of Comfort Management | From 1h before the date of life-support withdrawal to date of ICU discharge or death, whichever came first, assessed up to 28 days
  Proportion of patients with more than one gasp (≥ 2)
Assessment of Communication with Relatives | From inclusion to date of ICU discharge, assessed up to 28 days
  Proportion of relatives who had at least three meetings with ICU caregivers
Assessment of Communication with Relatives | From inclusion to date of ICU discharge, assessed up to 28 days
  Proportion of meetings conducted jointly by a senior physician and a nurse
Assessment of Communication with Relatives | From inclusion to date of ICU discharge, assessed up to 28 days
  Proportion of relatives who had a meeting with a psychologist
Assessment of Conflicts | From inclusion to date of ICU discharge, assessed up to 28 days
  Level of conflicts between ICU healthcare givers and relatives, as rated on a 0-10 Likert scale. A higher score indicates a more intense conflict.
Assessment of Conflicts | From inclusion to date of ICU discharge, assessed up to 28 days
  Level of conflicts between among healthcare professionals, as rated on a 0-10 Likert scale. A higher score indicates a more intense conflict.
Assessment of Conflicts | From inclusion to date of ICU discharge, assessed up to 28 days
  Level of conflicts between among relatives, as rated on a 0-10 Likert scale. A higher score indicates a more intense conflict.
Assessment of Quality of Dying by Relatives | From inclusion to 1 month after death of the patient
  Quality of Dying and Death questionnaire (QODD-1) assessed 1 month after death, as rated on a 0-10 Likert scale. Higher scores correlate with a more satisfactory level of care.
Anxiety and Depression in Relatives | From inclusion to 1, 3, 6, and 12 months after the death of the patient
  Hospital Anxiety and Depression Scale (HADS) assessed 1, 3, 6, and 12 months after death. HADS min = 0, max = 42; Higher scores correlate with increased risk of anxiety and depression.
Post-Traumatic Stress Disorders in Relatives | From inclusion to 1, 3, 6, and 12 months after the death of the patient
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) assessed 1, 3, 6, and 12 months after death. PCL-5 min = 0, max = 80; Higher scores correlate with increased risk of posttraumatic stress.
Prolonged Grief in Relatives | From inclusion to 12 months after the death of the patient
  Prolonged Grief Disorder scale (PG-13) assessed 12 months after death. PG-13 min = 4, max = 48; Higher scores correlate with increased risk of prolonged grief.
Assessment of Quality of Dying by Healthcare Professionals | After the death of the patient, assessed up to 28 days
  Quality of Dying and Death questionnaire (QODD-1), as rated on a 0-10 Likert scale. Higher scores correlate with a more satisfactory level of care.
Psychological Impact on Healthcare Professionals | After the death of the patient, assessed up to 28 days
  Measure of Moral Distress for Healthcare Professionals (MMD-HP). MMD-HP min = 0, max = 432; Higher scores correlate with increased risk of moral distress.
Impact on ICU Organization and Staff | Up to 2 years
  Perceived Stressors in Intensive Care Units (PS-ICU) assessing burnout at the end of the inclusion period. PS-ICU min = 0, max = 104; Higher scores correlate with increased risk of stress at work.
Impact on ICU Organization and Staff | Up to 2 years
  Maslach Burnout Inventory (MBI) assessing burnout at the end of the inclusion period. MBI min = 0, max = 132; Higher scores correlate with increased risk of burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Amélie SEGUIN, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 2027
Access Criteria: Open access